CLINICAL TRIAL: NCT06967610
Title: Phase II Study of Combined Pirtobrutinib, Venetoclax and Obinutuzumab (PVO) Time-limited Treatment for Patients With Recurrent Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL).
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0271; NCI-2025-03338 (Other: NCI-CTRP Clinical Registry")
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Leukemia (SLL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — pirtobrutinib; venetoclax; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- V-Exposed (Experimental): Venetoclax Exposed: Treatment with Pirtobrutinib+Venetoclax+Obinutuzumab Q4W
  Interventions: Drug: Pirtobrutinib; Drug: Venetoclax; Drug: Obinutuzumab
- V-Naive (Experimental): Venetoclax Naive: Treatment with Pirtobrutinib+Venetoclax+Obinutuzumab Q4W
  Interventions: Drug: Pirtobrutinib; Drug: Venetoclax; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Pirtobrutinib — Given PO 200mg daily
Drug: Venetoclax — Given PO daily
Drug: Obinutuzumab — Given IV 100mg day 1, 900 mg day 2, 100mg days 8, 15

SUMMARY:
To learn if the drug combination pirtobrutinib, venetoclax, and obinutuzumab can help to control relapsed CLL/SLL.

DETAILED DESCRIPTION:
Primary Objective:

- Rate of bone marrow undetectable Measurable Residual Disease (10-4 sensitivity; uMRD4) at end of Cycle 13.

Secondary Objectives:

* Blood uMRD6 rate at end of cycles 9, 13, 19, 25.
* 2018 iwCLL response rates defined as complete response (CR), CR with incomplete count recovery (CRi), partial response (PR), overall response (OR), stable disease (SD), and progressive disease (PD) at cycle 13.
* Progression-free (PFS) and overall survival (OS); time to blood uMRD6 relapse; safety and tolerability.

ELIGIBILITY:
Eligibility Criteria:

1. Age 18 years or older.
2. Diagnosis of CLL/SLL per 2018 iwCLL criteria (See Appendix 1).
3. Participants with previously treated CLL requiring therapy based on 2018 iwCLL criteria.
4. The participant is able to take oral medications.
5. Willing and capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.
6. Prior or ongoing therapy with covalent BTKi is allowed, but not required.
7. Prior or ongoing therapy (at least for six months) with BCL2i is allowed, but not required. Prior therapy with combined BTKi and BCL2i or triplet BTKi, BCL2 and anti-CD20 mAb is allowed, but Participants need to be at least six months after completion of combination therapy. Participants with history of prior venetoclax therapy should have achieved at least a partial response or better while receiving venetoclax therapy.
8. Participants are required to have the following washout periods prior to planned Cycle 1 Day1 (C1D1).

   * Targeted agents, investigational agents, therapeutic monoclonal antibodies or cytotoxic chemotherapy: 5 half-lives or 2 weeks, whichever is shorter
   * immunoconjugated antibody treatment within 10 weeks
   * broad field radiation (≥ 30% of the bone marrow or whole brain radiotherapy) must be completed 14 days prior to enrollment
   * palliative limited field radiation must be completed 7 days prior to enrollment
9. Prior treatment-related AEs must have recovered to Grade ≤ 1 with the exception of alopecia and Grade 2 peripheral neuropathy.
10. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2.
11. Participants must have adequate renal and hepatic function:

    * Serum bilirubin ≤1.5 x upper limit of normal (ULN) or ≤3 x ULN for Participants with Gilbert's disease or disease involvement by CLL/SLL.
    * Serum creatinine clearance of ≥30ml/min (calculated or measured).
    * ALT and AST ≤3.0 x ULN, unless clearly due to documented disease involvement, in which case ALT and AST ≤5.0 x ULN
12. Adequate bone marrow function:

    * Platelet count of ≥50,000/μl, with no platelet transfusion in prior 2 weeks.
    * ANC ≥750/μl in the absence of growth factor support within 7 days of screening assessment.
    * Hemoglobin ≥8g/dL, independent of transfusions within 7 days of screening assessment. Please refer to Appendix 4 for details of adjustments of toxicities in participants with abnormal baseline values)
13. Adequate coagulation, defined as activated partial thromboplastin time (aPTT) or partial thromboplastin time and prothrombin time (PT) or international normalized ratio (INR) not greater than 1.5 x ULN.
14. Women of childbearing potential must have a negative serum beta human chorionic gonadotropin (β-hCG) pregnancy test result at the time of screening and serum or urine β-hCG pregnancy test within 7 days prior to the first dose of study drugs and must agree to use both a highly effective method of birth control (eg, implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], complete abstinence, or sterilized partner) and a barrier method (eg., condoms, vaginal ring, sponge, etc) during the period of therapy and for 6 months after the last dose of study drug (pirtobrutinib and Obinutuzumab) and 12 months after the last dose of obinutuzumab. Women of nonchildbearing potential are those who are postmenopausal (defined as absence of menses for ≥1 year) or who have had a bilateral tubal ligation or hysterectomy. Men who have partners of childbearing potential must agree to use effective contraception, defined above, during the study and for 30 days following the last dose of study drug

Exclusion Criteria:

1. Participants who experienced progression of disease according to 2018 iwCLL criteria while on venetoclax will be excluded.
2. Patient with prior history of Richter's syndrome or current Richter's Syndrome.
3. Participants with known hypersensitivity to any of the excipients of pirtobrutinib, venetoclax,obinutuzumab or to any intended study medications.
4. Known or suspected history of central nervous system (CNS) involvement by CLL/SLL.
5. History of bleeding diathesis.
6. Participants who experienced a major bleeding event on a prior BTK inhibitor.• NOTE: Major bleeding is defined as bleeding having one or more of the following features: life-threatening bleeding with signs or symptoms of hemodynamic compromise; bleeding associated with a decrease in the hemoglobin level of at least 2 g/dL; or bleeding in a critical area or organ (e.g., retroperitoneal, intraarticular, pericardial, epidural, or intracranial bleeding or intramuscular bleeding with compartment syndrome).
7. History of stroke or intracranial hemorrhage within 6 months of enrollment.
8. Participants requiring therapeutic anticoagulation with warfarin or another vitamin K antagonists.
9. Major surgery within 4 weeks of planned start of study therapy.
10. A significant history of renal, neurologic, psychiatric, endocrine, metabolic or immunologic disorder, that, in the opinion of the Investigator, would adversely affect the participant's participation in this study or interpretation of study outcomes.
11. History of allogeneic or autologous stem cell transplant (SCT) or chimeric antigen receptor-modified Tcell (CAR-T) therapy within 60 days of enrollment or presence of any of the following, regardless of prior SCT and/or CAR-T therapy timing:

    * active graft versus host disease (GVHD);
    * cytopenia from incomplete blood cell count recovery post-transplant;
    * need for anti-cytokine therapy for toxicity from CAR-T therapy; residual symptoms of neurotoxicity > Grade 1 from CAR-T therapy;
    * ongoing immunosuppressive therapy (> 20 mg prednisone or equivalent daily).
12. Active uncontrolled auto-immune cytopenia (e.g., autoimmune hemolytic anemia [AIHA], idiopathic thrombocytopenic purpura [ITP]) for which new therapy was introduced or existing therapy was escalated within the 4 weeks prior to study enrollment to maintain adequate blood counts.
13. Participants who experienced grade >3 arrhythmia on prior treatment with BTK inhibitor.
14. Significant cardiovascular disease, defined as any of the following:

    1. Unstable angina or acute coronary syndrome within the past 2 months.
    2. History of myocardial infarction within 6 months prior to planned start of study treatment.
    3. Documented left ventricular ejection fraction (LVEF) by any method of ≤ 45% in the 12 months prior to planned start of study treatment.
    4. ≥ Grade 3 New York Heart Association (NYHA) functional classification system of heart failure.
    5. uncontrolled or symptomatic arrhythmias
15. Prolongation of the QT interval corrected (QTc - see Appendix 3) for heart rate using Fredericia's Formula (QTcF) > 470 msec on an EKG during screening.

    1. QTcF is calculated using Fredericia's Formula (QTcF = QT/(RR^0.33)
    2. Correction of suspected drug-induced QTcF prolongation or prolongation due to electrolyte abnormalities can be attempted at the Investigator's discretion, and only if clinically safe to do so with either discontinuation of the offending drug or switch to another drug not known to be associated with QTcF prolongation or electrolyte supplementation.
    3. Correction of QTc for underlying bundle branch block (BBB) permissible. Participants with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker
16. Hepatitis B or hepatitis C testing indicating active/ongoing infection based on screening laboratory tests as defined as:

    1. Hepatitis B virus (HBV): Participants with positive hepatitis B surface antigen (HBsAg) are excluded. Participants with positive hepatitis B core antibody (anti-HBc) and negative HBsAg require hepatitis B polymerase chain reaction (PCR) evaluation. Participants who are hepatitis B PCR positive will be excluded.
    2. Hepatitis C virus (HCV): positive hepatitis C antibody. If positive hepatitis C antibody result, participant will need to have a negative result for hepatitis C ribonucleic acid (RNA) . Participants who are hepatitis C RNA positive will be excluded.
17. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to, uncontrolled systemic infection (viral, bacterial, parasitic or fungal) or other clinically significant active disease process which in the opinion of the Principal Investigator may pose a risk for patient participation. Screening for chronic conditions is not required.
18. Known Human Immunodeficiency Virus (HIV) infection, regardless of CD4 count. For participants with unknown HIV status, HIV testing will be performed at screening and result must be negative for enrollment.
19. Known active CMV infection. Participants with unknown or negative status are eligible.
20. Vaccination with live vaccine within 28 days prior to enrollment
21. Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal (GI) absorption of the oral administered study treatments.
22. Active other malignancy unless in remission and with life expectancy > 2 years. with exception of participants diagnosed with basal cell or squamous cell carcinoma of the skin or carcinoma "in situ" of the cervix or breast who are eligible even if diagnosed within 2 years. If Participants have another malignancy that was treated within the last 2 years, such participants may be enrolled, if the likelihood of requiring systemic therapy for this other malignancy within 2 years is less than 10%, as determined by an expert in that particular malignancy at MD Anderson Cancer Center, and after consultation with the Principal Investigator.
23. Current treatment with strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers. A washout period of at least 5 half-lives of these agents following discontinuation before study entry is required (treatment with moderate CYP3A4 inhibitors or inducers is not excluded). Because of their effect on CYP3A4, use of any of the following within 7 days of study therapy start or planned use during study participation is prohibited i. Grapefruit or grapefruit products ii. Seville oranges or products from Seville oranges iii. Star fruit.
24. Current treatment with the following P-gp inhibitors: amiodarone, clarithromycin, cyclosporine, erythromycin, ketoconazole, and verapamil. A washout period of at least 5 half-lives of the inhibitor before study entry is required.
25. Participants that are pregnant or plan to become pregnant during the study or within 1 month of the last dose of study treatment.

25) Participants that are lactating or plan to breastfeed during the study or within 1 week of the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2031-06-01 (Estimated); Study Completion 2033-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferrajoli, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org